CLINICAL TRIAL: NCT00913692
Title: A Randomized Double-Blind Control-Comparison Crossover Trial of Oral Glutamine to Suppress Frequently Recurrent Herpes Labialis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow recruitment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jeffrey Cohen, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 090159; 09-I-0159
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Herpes Labialis; Herpes Simplex Virus
Keywords: Glutamine; Herpes Labialis; Herpes Simplex Virus; Cold Sore
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex | interventions — Glutamine; Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Glutamine — Subjects were randomized to take one of the study agents, 15 gm by mouth twice daily for 5 months. After a 2 week washout period, subjects began the other agent at 15 gm by mouth twice daily for 5 months.
Drug: Glycine — Subjects were randomized to take one of the study agents, 15 gm by mouth twice daily for 5 months. After a 2 week washout period, subjects began the other agent at 15 gm by mouth twice daily for 5 months.

SUMMARY:
Background:

* A cold sore is usually a blistering rash on or near the lips, caused by infection with herpes simplex virus. After the first infection, the virus goes into a dormant (inactive) state, but it can continue to cause cold sores.
* Most people with the herpes simplex virus have a few episodes of cold sores per year. However, some individuals may have many recurrent episodes that are uncomfortable and may cause embarrassment. Researchers are attempting to find treatments that can decrease the number of cold sore episodes for people who have six or more episodes per year.
* Glutamine is a molecule called an amino acid and is one of the components that make up proteins in the body. Clinical studies using glutamine have addressed the potential of glutamine to improve immune function and to heal damaged tissue or to help healing.

Objectives:

- To find out if the dietary supplement glutamine can help individuals with frequently recurring (more than six episodes per year) cold sores.

Eligibility:

* Patients between 18 and 65 years of age who have a history of having six or more cold sore episodes per year, and have not received certain kinds of drug treatment for the cold sores within 1 month of beginning the study.
* Patients who have two or more episodes of cold sores caused by the herpes simplex virus will be eligible for treatment as part of this study.

Design:

* Initial clinical visit for a physical examination and medical history, at which blood samples will be drawn for testing.
* Eligible participants will undergo a 4-month screening period. Patients who develop sores during this period will visit the NIH to have the sore examined to determine if it is caused by the herpes virus. Patients who have two or more episodes of cold sores caused by the herpes simplex virus will be eligible for treatment.
* Patients who are eligible for treatment will provide an initial blood sample and will receive randomized doses of either glutamine or glycine (another amino acid), which must be taken on a regular schedule twice daily, mixed with either liquid or soft food. Patients who develop sores during this period will visit the NIH to have the sore examined to determine if it is caused by the herpes virus. Blood, urine, and saliva specimens will be collected each month during the treatment period. A 2-week washout period will occur between the 2 treatment periods when no doses of glutamine or glycine will be taken.
* Patients will then undergo a second 5-month treatment period with either glutamine or glycine (whichever was not given in the first part of the study), taken in the same manner as before. Patients who develop sores during this period will visit the NIH to have the sore examined to determine if it is caused by the herpes virus.
* After the second treatment, patients will remain in touch with researchers for 1 month to note any changes.

DETAILED DESCRIPTION:
Frequently recurrent herpes simplex virus type 1 (HSV-1) infection of the lips or perioral area, known as herpes labialis, or commonly as cold sores, can cause discomfort, pain, and embarrassment. Traditional antiviral therapies are moderately effective in suppressing these recurrences. Studies have shown that the amino acid glutamine can affect HSV-1 reactivation in vitro. Glutamine has been studied in various clinical situations and has been found to decrease morbidity in critically ill patients (reducing nosocomial infections), in patients receiving chemotherapy or undergoing bone marrow transplantation (reducing severity of stomatitis, reducing incidence of infection, shortening hospital stay), and in patients with short gut syndrome (decreasing requirement for parenteral nutrition). No significant adverse consequences of glutamine therapy have been reported in these patients. We will conduct a randomized, double-blind, control-comparison crossover trial comparing the efficacy of glutamine versus glycine (control) to suppress recurrences of herpes labialis in patients with frequent episodes (greater than or equal to 6 per year). Based on our in vitro and in vivo data, we hypothesize that oral glutamine will decrease the number of recurrences of herpes labialis during a 5-month treatment period in participants with frequently recurring herpes labialis compared with control.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults, ages 18 to 65, who report a history of 6 or more episodes of herpes labialis per year.
  2. Subject agrees to refrain from using over the counter (OTC), prescription or supplemental antiviral medications without obtaining permission from the study team during the course of the study.
  3. Women with child-bearing potential are required and willing to practice two effective methods of birth control beginning with the first treatment period and continuing until the end of the study.
  4. Women with child-bearing potential are required to have a negative pregnancy test at the time of enrollment and at the time of randomization.
  5. To be eligible for randomization in the treatment phase of the study, the participants must experience at least 2 clinically confirmed episodes of herpes labialis, 1 of which must be virologically confirmed, during the 4 month screening period.

EXCLUSION CRITERIA:

1. Oral or intravenous antiviral therapy < 4 weeks before enrollment or during the study with the following agents is not permitted: acyclovir (intravenous), ganciclovir (intravenous or oral), valganiciclovir (oral), cidofovir (intravenous), or foscarnet (intravenous).

   1. Suppressive therapy with oral acyclovir, valacyclovir or famciclovir or with topical antivirals 4 weeks prior to enrollment or during the study is not permitted.
   2. Use of oral acyclovir or valacyclovir or famciclovir or topical antiviral ointments or creams for the treatment of herpes labialis outbreaks during the study is permitted AFTER the outbreak has been documented by the study team..
2. Evidence of active herpes labialis reactivation at the time of enrollment. The volunteer can be enrolled after resolution of herpes labialis and if inclusion and exclusion criteria are still met.
3. Subjects with conditions associated with immunodeficiency (e.g., human immunodeficiency virus infection) or conditions requiring either daily systemic corticosteroids exceeding a dose equivalent to10 mg/day of prednisone or other significant immunosuppressant therapy (e.g., organ or stem cell transplantation).
4. Persons with significant liver or kidney disease [serum glutamic oxaloacetic transaminase [SGOT], serum glutamine pyruvic transaminase [SGPT], or alkaline phosphatase > 2.5 times the upper limit of normal (ULN), total bilirubin > 1.5 times the ULN, or serum creatinine > 1.5 times the ULN].
5. Persons with an active seizure disorder. For persons with prior history of seizures, the person should be seizure free for 5 years and not on any anti-seizure medication in order to be enrolled into the study. (Since glutamine is metabolized to glutamate and ammonia, and glutamate is the main excitatory neurotransmitter in the central nervous system (CNS), there is a theoretical increased risk of seizures).
6. Women who are known to be pregnant (pregnancy category C) or breastfeeding (it is not known whether glutamine is excreted in human milk).
7. History of allergic reaction to glutamine or glutamic acid or their derivatives (e.g., monosodium glutamate) or to glycine or sucralose.
8. Subjects cannot take supplemental amino acids (e.g., glutamine, glycine, arginine, other amino acids) or high protein supplements, such as Boost within 30 days of enrollment into the study or during the study (except for study drug amino acid). Subjects can take vitamins.
9. Persons treated with atypical neuroleptics such as clozapine (Clozaril, FazoCIo) or olanzapine (Zyprexa, Zydis).
10. Participation in any study involving investigational drugs within 30 days prior to entry into this trial.
11. Any condition (e.g., schizophrenia, psychosis, major depression, mental deficiency or illness) or major co-morbidity that the study investigator thinks might compromise the person's ability to comply with the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson PM, Ramsay NK, Shu XO, Rydholm N, Rogosheske J, Nicklow R, Weisdorf DJ, Skubitz KM. Effect of low-dose oral glutamine on painful stomatitis during bone marrow transplantation. Bone Marrow Transplant. 1998 Aug;22(4):339-44. doi: 10.1038/sj.bmt.1701317. PMID 9722068
- [Background] Aquino VM, Harvey AR, Garvin JH, Godder KT, Nieder ML, Adams RH, Jackson GB, Sandler ES. A double-blind randomized placebo-controlled study of oral glutamine in the prevention of mucositis in children undergoing hematopoietic stem cell transplantation: a pediatric blood and marrow transplant consortium study. Bone Marrow Transplant. 2005 Oct;36(7):611-6. doi: 10.1038/sj.bmt.1705084. PMID 16086046
- [Background] Baker D, Eisen D. Valacyclovir for prevention of recurrent herpes labialis: 2 double-blind, placebo-controlled studies. Cutis. 2003 Mar;71(3):239-42. PMID 12661753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November 2009 at the NIH Clinical Center outpatient clinic. Eleven study participants were enrolled and screened from 11/2009 - 11/2010. Two of these participants proceeded to the treatment phase of the study.
Pre-assignment Details: Participants were enrolled and randomized to the treatment phase only if they met the eligibility criteria after completing the 4 month screening phase. After completion of phase 1 of treatment, there was a 2 week wash out period before beginning phase 2 of treatment.
Groups:
- Glutamine (Study Agent) or Glycine (Placebo): Participants were enrolled and monitored to document presence of 2 clinically confirmed episodes of herpes labialis, 1 of which must be virologically confirmed, during the screening period. Participants took 15 gm of study agent or placebo by mouth twice daily for 5 months followed by a 2 week wash-out. Then participants took the other agent for another 5 months.
Period: Screening (4 Months)
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Started | 11
Completed | 2
Not Completed | 9
Not completed — Physician Decision | 3
Not completed — Not eligible after screening phase. | 6
Period: Treatment Phase 1 (5 Months)
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Physician Decision | 1
Period: Washout (2 Weeks)
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Started | 1
Completed | 1
Not Completed | 0
Period: Treatment Phase 2 (5 Months)
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Does Oral Glutamine Reduce the Number of Recurrences of Herpes Labialis, Diagnosed by Clinical and Microbiologic Criteria, in Healthy Participants With Frequently Recurrent Disease.
Description: During all phases of the study, participants returned to clinic whenever they had a herpes labialis outbreak for staff to assess, obtain a viral swab and document. If unable to return to clinic in the time frame specified in the protocol, participants would take a photo and obtain a swab of the lesion. The number of outbreaks would be measured during each phase.
Time Frame: The screening phase time frame was 4 months. Treatment phase 1 was 5 months. Washout phase was 2 weeks. Treatment phase 2 was 5 months.
Population: One participant completed the study and one participant started the 1st treatment phase, but was withdrawn during the first treatment phase, hence the primary outcome could not be measured and analyzed.
Measure: Number; unit: herpes labialis lesions
Groups:
- Glutamine (Study Agent) or Glycine (Placebo): One participant completed the study and one participant started the 1st treatment phase, but was withdrawn during the first treatment phase, hence the primary outcome could not be measured and analyzed.
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 0

2. Secondary Outcome: Does Oral Glutamine Reduce the Number of Clinical Recurrences of Herpes Labialis With or Without PCR Confirmation?
Description: During all phases of the study, participants returned to clinic whenever they had a herpes labialis outbreak for staff to assess, obtain a viral swab and document. If unable to return to clinic in the time frame specified in the protocol, participants would take a photo and obtain a swab of the lesion. The number of recurrences would be documented during each phase of the study.
Time Frame: as for outcome 1
Population: One participant completed the study and one participant started the 1st treatment phase, but was withdrawn during the first treatment phase, hence the secondary outcomes could not be measured and analyzed.
Measure: Median (Standard Deviation); unit: herpes labialis lesions
Groups:
- Glutamine (Study Agent) or Glycine (Placebo): One participant completed the study and one participant started the 1st treatment phase, but was withdrawn during the first treatment phase, hence the secondary outcomes could not be measured and analyzed.
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 0

3. Secondary Outcome: Does Oral Glutamine Reduce the Time to First Recurrence of Herpes Labialis Diagnosed by Clinical and Microbiologic Criteria or Diagnosed by Clinical Criteria With or Without PCR Confirmation?
Description: During all phases of the study, participants returned to clinic whenever they had a herpes labialis outbreak for staff to assess, obtain a viral swab and document. If unable to return to clinic in the time frame specified in the protocol, participants would take a photo and obtain a swab of the lesion. The number of recurrences and start and end dates of each recurrence would be documented during each phase of the study.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: days
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 0

4. Secondary Outcome: Does Oral Glutamine Reduce the Duration of Recurrences?
Description: During all phases of the study, participants returned to clinic whenever they had a herpes labialis outbreak for staff to assess, obtain a viral swab and document. If unable to return to clinic in the time frame specified in the protocol, participants would take a photo and obtain a swab of the lesion. The number of recurrences and start and end dates of each recurrence would be documented.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: days
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 0

5. Secondary Outcome: Does Oral Glutamine Reduce the Area of Recurrent Lesions?
Description: During all phases of the study, participants returned to clinic whenever they had a herpes labialis outbreak for staff to assess, obtain a viral swab and document. If unable to return to clinic in the time frame specified in the protocol, participants would take a photo and obtain a swab of the lesion. The number of recurrences, start and end dates of each recurrence and measurement of each lesion during each phase of the study would be documented.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mm squared
Arm/Group | Glutamine (Study Agent) or Glycine (Placebo)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of drug to 1 month after the last dose of drug. Serious adverse events (SAEs) and non-serious adverse events (AEs) were followed until resolution or until the AE/SAE has stabilized and no more follow-up is required.
Groups:
- Treatment Phase 1; Washout; Treatment Phase 2: 2 participants were eligible for the treatment phase of the study after the screening period. 1 participant completed treatment phase 1 & 2. 1 participant was withdrawn from treatment phase 1 after the investigator decided to place the study on hold.
Arm/Group | Treatment Phase 1 | Washout | Treatment Phase 2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase 1 (N=2) | Washout (N=1) | Treatment Phase 2 (N=1)
abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (3) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) — pitting edema to bilateral lower legs and ankles
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — elevated AST
Blood lactate dehydrogenase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) — elevated LDH
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tension Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — bizarre dreams
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The protocol was terminated early due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No